CLINICAL TRIAL: NCT04309916
Title: A Multicenter, Double-blind, Randomized, Active-controlled Phase 4 (Pilot) Study to Evaluate the Efficacy and Safety of Tegoprazan in ERD Patients With Nighttime Heartburn and Sleep Disturbance
Brief Title: Study to Evaluate the Efficacy and Safety of Tegoprazan in ERD Patients With Nighttime Heartburn and Sleep Disturbance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KCAB_002
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Erosive Reflux Disease
MeSH Terms: interventions — tegoprazan; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tegoprazan 50mg (Experimental): Tegoprazan 50mg tablet, once daily, oral administration
  Interventions: Drug: Tegoprazan
- Esomeprazole 40mg (Active Comparator): Esomeprazole 40mg tablet, once daily, oral administration
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Tegoprazan — Tegoprazan 50mg tablet
  Arms: Tegoprazan 50mg
Drug: Esomeprazole — Esomeprazole 40mg tablet
  Arms: Esomeprazole 40mg

SUMMARY:
This study aims to compare the nighttime heartburn and sleep disturbance improvement effect of Tegoprazan 50mg and Eomeprazole 40mg in patients with ERD patients.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized, active-controlled phase 4 (pilot) study. Subjects will be randomly assigned to one of the two treatment groups (tegoprazan 50mg, esomeprazole 40mg)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 19 and 75 years
2. Subjects who have erosive reflux disease

Exclusion Criteria:

1. Unable to undergo upper GI endoscopy
2. Symptoms of primary or secondary esophageal movement disorders
3. Planning or Perform surgery that can affect gastric acid secretion (e.g., upper gastrectomy, Vagotomy, etc.)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Time to first nighttime heartburn-free interval (days)) | 2 week
  Number of days to reach the without symptoms of nighttime heartburn after the start of drug administration for clinical trials.

SECONDARY OUTCOMES:
Percentage of days without nighttime heartburn during the 2-week dosing period | 2 week
  Percentage of days without nighttime heartburn = Number of days without nighttime heartburn symptoms during the dosing period / Number of days when nighttime heartburn was assessed x 100

CONTACTS AND LOCATIONS:
Overall Officials: Sang Kil Lee, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea